CLINICAL TRIAL: NCT01553279
Title: A Phase III Open-label Randomised Study, to Evaluate the Immunogenicity and Safety of the Concomitant Administration of V419 (PR5I) Given at 2, 3 and 4 Months of Age With Two Types of Meningococcal Serogroup C Conjugate (MCC) Vaccines Given at 3 and 4 Months of Age, and Followed by the Administration at 12 Months of Age of a Combined Haemophilus Influenzae Type b-MCC Vaccine
Brief Title: Immunogenicity and Safety of V419 (PR51) in Combination With MCC in Infants and Toddlers (V419-011)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MCM Vaccines B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V419-011; 2011-002413-11 (EudraCT Number); PRI01C (Other: MCMVaccBV Protocol ID); V419-011 (Other: Merck Protocol Number)
Record Dates: First submitted 2012-03-07; First posted 2012-03-14 (Estimated); Results first posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Neisseria Meningitidis; Bacterial Infections; Virus Diseases
MeSH Terms: conditions — Bacterial Infections; Virus Diseases | interventions — Vaxelis; 13-valent pneumococcal vaccine; Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- V419 and MCC-TT (Experimental): Participants received 3 doses of V419 (at 2, 3, and 4 months of age) and 2 doses of MCC-TT (at 3 and 4 months of age), followed by a single dose of Hib-MCC at 12 months of age. As routine vaccination, participants also received 2 doses of Prevnar 13® (at 2 and 4 months of age) and 1 dose of a measles, mumps, and rubella (MMR) vaccine (at 12 months of age).
  Interventions: Biological: V419; Biological: PREVNAR 13®; Biological: MCC-TT; Biological: Hib-MCC; Biological: MMR Vaccine
- V419 and MCC-CRM (Experimental): Participants received 3 doses of V419 (at 2, 3, and 4 months of age) and 2 doses of MCC-CRM (at 3 and 4 months of age), followed by a single dose of Hib-MCC at 12 months of age. As routine vaccination, participants also received 2 doses of Prevnar 13® (at 2 and 4 months of age) and 1 dose of an MMR vaccine (at 12 months of age).
  Interventions: Biological: V419; Biological: PREVNAR 13®; Biological: MCC-CRM; Biological: Hib-MCC; Biological: MMR Vaccine

INTERVENTIONS:
Biological: V419 — Diphtheria and Tetanus toxoids and acellular Pertussis adsorbed, inactivated Poliovirus, Haemophilus b conjugate [meningococcal outer membrane protein complex], and Hepatitis B [recombinant] vaccine administered via 0.5 mL intramuscular injection.
  Other Names: PR51, VAXELIS®
Biological: PREVNAR 13® — Pneumococcal conjugate vaccine (13-valent, adsorbed) administered via 0.5 mL intramuscular injection (routine vaccination).
Biological: MCC-TT — Meningococcal Group C polysaccharide conjugate vaccine to tetanus toxoid adsorbed 0.5 mL intramuscular injection at 3 and 4 months of age
  Other Names: NEISVAC-C®
  Arms: V419 and MCC-TT
Biological: MCC-CRM — Meningococcal Group C conjugate vaccine to CRM-197 adsorbed 0.5 mL intramuscular injection at 3 and 4 months of age
  Other Names: MENJUGATE®
  Arms: V419 and MCC-CRM
Biological: Hib-MCC — Haemophilus type b and meningococcal Group C conjugate vaccine administered via 0.5 mL intramuscular injection.
  Other Names: MENITORIX®
Biological: MMR Vaccine — Measles, mumps, and rubella vaccine (live) given via 0.5 mL intramuscular injection (routine vaccination).
  Other Names: M-M-RVAXPRO®

SUMMARY:
The primary objectives of this study are to evaluate the immunogenicity and safety of concomitant administration of V419 (PR51) with 2 types of meningococcal serogroup C conjugate (MCC) vaccines to healthy infants at 3 and 4 months of age in terms of antibody seroprotection rate (SPR) to MCC. Participants also received a Haemophilus influenza type B (Hib)-MCC vaccination at 12 months of age. It was hypothesized that the SPR to MCC at 1 month post-dose 2 of either tetanus toxoid conjugated Meningo C (MCC-TT) or CRM197 conjugated Meningo C (MCC-CRM) vaccines would be acceptable when administered concomitantly with V419.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infant 46 to 74 days of age (both inclusive)
* Parent(s)/legal representative able to comply will the study procedures

Exclusion Criteria:

* Is participating in a study with an investigational compound or device since birth
* Has a history of congenital or acquired immunodeficiency
* Has a history of leukemia, lymphoma, malignant melanoma or myeloproliferative disorder
* Has a chronic illness that could interfere with study conduct or completion
* Has hypersensitivity to any of the vaccines components or history of a life-threatening reaction to a vaccine containing the same substances as the study vaccines or contraindication to any of the study vaccines
* Has a history, or mother has a history, of hepatitis B virus surface antigen (HBsAg) seropositivity
* Has a coagulation disorder that contraindicate intramuscular injection
* Has a history of vaccination with a hepatitis B, Haemophilus influenzae type b conjugate, diphtheria, tetanus, pertussis (acellular or whole-cell), poliovirus, pneumococcal conjugate or polysaccharide, meningococcal serogroup C conjugate, measles, mumps, or rubella containing vaccine(s)
* Has a history of hepatitis B, Haemophilus influenzae type b, diphtheria, tetanus, pertussis, poliomyelitis, invasive pneumococcal, meningococcal serogroup C, measles, mumps or rubella infection
* Has received immune globulin, blood or blood-derived products, immunosuppressive agents systemic corticosteroids since birth
* Has received vaccination with an inactivated (except influenza vaccine) or conjugated or live vaccine in the last 30 days or vaccination with an inactivated influenza vaccine in the last 14 days
* Has received antipyretic, analgesic and non-steroidal anti-inflammatory medications in the last 48 hours
* Has a febrile illness or body temperature ≥38.0°C in the last 24 hours

Ages: 46 Days to 74 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 284 (Actual)
Dates: Start 2012-03-30 (Actual); Primary Completion 2013-09-27 (Actual); Study Completion 2013-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infant participants were enrolled at 11 study sites in the United Kingdom.
Groups:
- V419 and MCC-TT: In Part 1, participants received 3 doses of V419 (at 2, 3, and 4 months of age) and 2 doses of MCC-TT (at 3 and 4 months of age). In Part 2, participants received a single dose of Hib-MCC at 12 months of age. As routine vaccination, participants also received 2 doses of Prevnar 13® (at 2 and 4 months of age) and 1 dose of an MMR vaccine (at 12 months of age).
- V419 and MCC-CRM: In Part 1, participants received 3 doses of V419 (at 2, 3, and 4 months of age) and 2 doses of MCC-CRM (at 3 and 4 months of age). In Part 2, participants received a single dose of Hib-MCC at 12 months of age. As routine vaccination, participants also received 2 doses of Prevnar 13® (at 2 and 4 months of age) and 1 dose of an MMR vaccine (at 12 months of age).
Period: Part 1 (Infant Vaccinations)
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Started (Number Randomized) | 142 | 142
Completed | 140 | 141
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Period: Interim Period
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Started | 140 | 141
Completed | 137 | 139
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Period: Period 2: Toddler Vaccinations
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Started | 137 | 139
Completed | 134 | 132
Not Completed | 3 | 7
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM | Total
Number analyzed (Participants) | 142 | 142 | 284
Age, Continuous [Mean (Standard Deviation); unit: Days] | 62.6 (6.7) | 61.6 (7.2) | 62.1 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 67 | 129
  Male | 80 | 75 | 155

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Anti-Meningococcal Serogroup C (Anti-MCC) Antibody (Ab) Titre ≥1:8 Dil One Month After MCC-TT or MCC-CRM (Part 1)
Description: The acceptability (i.e., percentage of participants with anti-MCC Ab titre ≥1:8 dil) of the seroprotection rate (SPR) to MCC was determined 1 month after MCC-TT or MCC-CRM Dose 2. The SPR was considered acceptable if the lower bound of the 2-sided 95% CI was >90%. Serum Ab levels were assayed using the Meningo C rabbit complement serum bactericidal Ab (rSBA) assay.
Time Frame: Month 5 (1 month after MCC-TT/MCC-CRM Dose 2)
Population: All randomized and treated participants with data available and who had no protocol violations that could interfere with results are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 121 | 109
Percentage of Participants | 100.0 [97.0 to 100.0] | 99.1 [95.0 to 100.0]

2. Secondary Outcome: Percentage of Participants With Anti-Polyribosylribitol Phosphate (Anti-PRP) Antibody (Ab) Titre ≥0.15 µg/mL One Month After V419 Dose 3 (Part 1)
Description: The acceptability (i.e., percentage of participants with anti-PRP Ab titre ≥0.15 µg/mL) of the seroprotection rate (SPR) to Haemophilus influenza type b (Hib) was determined 1 month after the third dose of V419 in participants also treated with MCC-TT or MCC-CRM. The pooled (i.e., all V419-treated participants) SPR was considered acceptable if the lower bound of the 2-sided 95% CI was >80%. Serum Ab levels were determined with radioimmunoassay (RIA).
Time Frame: Month 5 (1 month after V419 Dose 3)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- V419 + MCC-TT/MCC-CRM: In Part 1, participants received 3 doses of V419 (at 2, 3, and 4 months of age) and 2 doses of MCC-TT or MCC-CRM (at 3 and 4 months of age).
Arm/Group | V419 + MCC-TT/MCC-CRM
Number analyzed (Participants) | 175
Percentage of Participants | 98.9 [95.9 to 99.9]

3. Secondary Outcome: Percentage of Participants With Anti-Meningococcal Serogroup C (Anti-MCC) Antibody (Ab) Titre ≥1:8 Dil and ≥1:128 Dil One Month After MCC-TT or MCC-CRM Doses 1 and 2 (Part 1)
Description: The percentage of participants with anti-MCC Ab titres ≥1:8 dil and ≥1:128 dil 1 month after MCC-TT or MCC-CRM Doses 1 and 2 was determined in participants also treated with V419. Serum Ab levels were assayed using the Meningo C rabbit complement serum bactericidal Ab (rSBA) assay.
Time Frame: Month 4 and Month 5 (1 month after MCC-TT/MCC-CRM Doses 1 and 2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 121 | 109
Percentage of Participants
  Post-MCC Dose 1: % with ≥1:8 dil: number analyzed (Participants) | 102 | 84
  Post-MCC Dose 1: % with ≥1:8 dil | 100.0 [96.4 to 100.0] | 96.4 [89.9 to 99.3]
  Post-MCC Dose 1: % with ≥1:128 dil: number analyzed (Participants) | 102 | 84
  Post-MCC Dose 1: % with ≥1:128 dil | 98.0 [93.1 to 99.8] | 84.5 [75.0 to 91.5]
  Post-MCC Dose 2: % with ≥1:8 dil | 100.0 [97.0 to 100.0] | 99.1 [95.0 to 100.0]
  Post-MCC Dose 2: % with ≥1:128 dil | 99.2 [95.5 to 100.0] | 99.1 [95.0 to 100.0]

4. Secondary Outcome: Geometric Mean Titres (GMTs) for Meningococcal Serogroup C (MCC) One Month After MCC-TT or MCC-CRM Doses 1 and 2 (Part 1)
Description: Anti-MCC antibody GMTs were determined 1 month after MCC-TT or MCC-CRM Doses 1 and 2 in participants also treated with V419. Serum antibody levels were assayed using the Meningo C rabbit complement serum bactericidal antibody (rSBA) assay.
Time Frame: Month 4 and Month 5 (1 month after MCC-TT/MCC-CRM Doses 1 and 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 125 | 111
Titres
  Post-MCC Dose 1 anti-MCC GMTs | 1353 [1058.4 to 1729.6] | 285.0 [201.5 to 403.1]
  Post-MCC Dose 2 anti-MCC GMTs | 2024.7 [1689.8 to 2425.9] | 1077.4 [847.5 to 1369.8]

5. Secondary Outcome: Antibody (Ab) Response Rates for V114 Antigens One Month After V114 Dose 3 (Part 1)
Description: The percentage of participants meeting Ab response rates for V14 antigens was determined after V114 Dose 3. Antibody response rate criteria for Haemophilus influenza Type B (PRP); hepatitis B (HBsAg); diphtheria; tetanus; and polio types 1, 2, and 3 are shown in the rows below. The percentage of seroresponders to pertussis seroresponders (pertussis toxoid [PT]; filamentous haemagglutinin (FHA); fimbrae types 2 and 3 [FIM]; and pertactin [PRN]) was determined as 1) if pre-vaccination Ab concentration <lower limit of quantification (LLoQ) but post-vaccination Ab concentration ≥LLoQ; or 2) if pre-vaccination Ab concentration was ≥LLoQ but post-vaccination Ab concentration was ≥pre-immunization levels. Antibody titres were measured by RIA for PRP, enhanced chemiluminescence assay (ECi) for HBsAg, micrometabolic inhibition test (MIT) for diphtheria and poliovirus, and enzyme-linked immunosorbent assay (ELISA) for tetanus, PT, FHA, FIM, and PRN.
Time Frame: Month 5 (1 month after V419 Dose 3)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 125 | 111
Percentage of Participants
  Anti-PRP ≥0.15 µg/mL: number analyzed (Participants) | 93 | 82
  Anti-PRP ≥0.15 µg/mL | 97.8 [92.4 to 99.7] | 100.0 [95.6 to 100.0]
  Anti-HBsAG ≥10 mIU/mL: number analyzed (Participants) | 93 | 82
  Anti-HBsAG ≥10 mIU/mL | 96.8 [90.9 to 99.3] | 96.3 [89.7 to 99.2]
  Anti-Diptheria ≥0.01 IU/mL: number analyzed (Participants) | 125 | 104
  Anti-Diptheria ≥0.01 IU/mL | 100.0 [97.1 to 100.0] | 100.0 [96.5 to 100.0]
  Anti-Diptheria ≥0.1 IU/mL: number analyzed (Participants) | 125 | 104
  Anti-Diptheria ≥0.1 IU/mL | 68.0 [59.1 to 76.1] | 74.0 [64.5 to 82.1]
  Anti-Tetanus ≥0.01 IU/mL: number analyzed (Participants) | 122 | 105
  Anti-Tetanus ≥0.01 IU/mL | 100.0 [97.0 to 100.0] | 100.0 [96.5 to 100.0]
  Anti-Tetanus ≥0.1 IU/mL: number analyzed (Participants) | 122 | 105
  Anti-Tetanus ≥0.1 IU/mL | 100.0 [97.0 to 100.0] | 100.0 [96.5 to 100.0]
  Anti-PT seroresponse: number analyzed (Participants) | 100 | 75
  Anti-PT seroresponse | 99.0 [94.6 to 100.0] | 100.0 [95.2 to 100.0]
  Anti-FHA seroresponse: number analyzed (Participants) | 100 | 74
  Anti-FHA seroresponse | 91.0 [83.6 to 95.8] | 90.5 [81.5 to 96.1]
  Anti-PRN seroresponse: number analyzed (Participants) | 100 | 73
  Anti-PRN seroresponse | 95.0 [88.7 to 98.4] | 90.4 [81.2 to 96.1]
  Anti-FIM seroresponse: number analyzed (Participants) | 100 | 75
  Anti-FIM seroresponse | 96.0 [90.1 to 98.9] | 96.0 [88.8 to 99.2]
  Anti-Polio 1 ≥ 1:8 dil: number analyzed (Participants) | 114 | 95
  Anti-Polio 1 ≥ 1:8 dil | 100.0 [96.8 to 100.0] | 100.0 [96.2 to 100.0]
  Anti-Polio 2 ≥ 1:8 dil: number analyzed (Participants) | 106 | 89
  Anti-Polio 2 ≥ 1:8 dil | 100.0 [96.6 to 100.0] | 100.0 [95.9 to 100.0]
  Anti-Polio 3 ≥ 1:8 dil: number analyzed (Participants) | 90 | 74
  Anti-Polio 3 ≥ 1:8 dil | 100.0 [96.0 to 100.0] | 100.0 [95.1 to 100.0]

6. Secondary Outcome: Antibody (Ab) Geometic Mean Titres (GMTs) for Haemophilus Influenza Type B (Polyribosylribitol Phosphate [PRP]) One Month After V114 Dose 3 (Part 2)
Description: The GMTs for PRP Ab titres were determined for each arm. Antibody titres for PRP were measured by radioimmunoassay (RIA).
Time Frame: Month 5 (1 month after V419 Dose 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 125 | 111
µg/mL | 6.44 [4.7 to 8.83] | 8.21 [6.08 to 11.09]

7. Secondary Outcome: Antibody (Ab) Geometic Mean Titres (GMTs) for Hepatitis B Surface Antigen (HBsAg) One Month After V114 Dose 3 (Part 2)
Description: The GMTs for HBsAg Ab titres were determined for each arm. Antibody titres for HBsAg were measured by enhanced chemiluminescence (ECi) assay.
Time Frame: Month 5 (1 month after V419 Dose 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 125 | 111
mIU/mL | 195.1 [150.7 to 252.7] | 247.7 [186.3 to 329.3]

8. Secondary Outcome: Antibody (Ab) Geometic Mean Titres (GMTs) for Diptheria One Month After V114 Dose 3 (Part 2)
Description: The GMTs for diphtheria Ab titres were determined for each arm. Antibody titres for diptheria were measured by enhanced micrometabolic inhibition test (MIT).
Time Frame: Month 5 (1 month after V419 Dose 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 125 | 111
IU/mL | 0.198 [0.165 to 0.237] | 0.22 [0.181 to 0.268]

9. Secondary Outcome: Antibody (Ab) Geometic Mean Titres (GMTs) for Tetanus One Month After V114 Dose 3 (Part 2)
Description: The GMTs for tetanus Ab titres were determined for each arm. Antibody titres for tetanus were determined with enzyme-linked immunosorbent assay (ELISA).
Time Frame: Month 5 (1 month after V419 Dose 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 125 | 111
IU/mL | 1.03 [0.9 to 1.17] | 0.95 [0.82 to 1.1]

10. Secondary Outcome: Antibody (Ab) Geometic Mean Titres (GMTs) for Pertussis Toxoid (PT) One Month After V114 Dose 3 (Part 2)
Description: The GMTs for PT Ab titres were determined for each arm. Antibody titres for PT were measured with enzyme-linked immunosorbent assay (ELISA).
Time Frame: Month 5 (1 month after V419 Dose 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 125 | 111
EU/mL | 131.5 [117.2 to 147.6] | 133.3 [118.3 to 150.2]

11. Secondary Outcome: Antibody (Ab) Geometic Mean Titres (GMTs) for Filamentous Haemagglutinin (FHA) One Month After V114 Dose 3 (Part 2)
Description: The GMTs for FHA were determined for each arm. Antibody titres for FHA were measured by enhanced chemiluminescence (ECi) assay.
Time Frame: Month 5 (1 month after V419 Dose 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 125 | 111
EU/mL | 50.4 [44.8 to 56.6] | 50.1 [43.7 to 57.4]

12. Secondary Outcome: Antibody (Ab) Geometic Mean Titres (GMTs) for Pertactin (PRN) One Month After V114 Dose 3 (Part 2)
Description: The GMTs for PRN were determined for each arm. Antibody titres for PRN were measured by enhanced chemiluminescence (ECi) assay.
Time Frame: Month 5 (1 month after V419 Dose 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 125 | 111
EU/mL | 90.4 [73.2 to 111.7] | 106.8 [83.7 to 136.3]

13. Secondary Outcome: Antibody (Ab) Geometic Mean Titres (GMTs) for Fimbrae Types 2 and 3 (FIM) One Month After V114 Dose 3 (Part 2)
Description: The GMTs for FIM were determined for each arm. Antibody titres for FIM were measured by enhanced chemiluminescence (ECi) assay.
Time Frame: Month 5 (1 month after V419 Dose 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 125 | 111
EU/mL | 401.7 [339.4 to 475.5] | 441.7 [363.2 to 537.2]

14. Secondary Outcome: Antibody (Ab) Geometic Mean Titres (GMTs) for Polio Types 1, 2, and 3 One Month After V114 Dose 3 (Part 2)
Description: The GMTs for polio types 1, 2, and 3 were determined for each arm. Antibody titres for polio types 1, 2, and 3 were measured by micrometabolic inhibition test (MIT).
Time Frame: Month 5 (1 month after V419 Dose 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titre (1/dil)
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 125 | 111
titre (1/dil)
  Anti-Polio 1 GMT: number analyzed (Participants) | 114 | 95
  Anti-Polio 1 GMT | 214 [164.9 to 277.7] | 257.9 [193.8 to 343.1]
  Anti-Polio 2 GMT: number analyzed (Participants) | 106 | 89
  Anti-Polio 2 GMT | 385.2 [288.2 to 514.9] | 400.6 [290.6 to 552.3]
  Anti-Polio 3 GMT: number analyzed (Participants) | 90 | 74
  Anti-Polio 3 GMT | 502.2 [370.2 to 681.4] | 405.1 [284.9 to 576]

15. Secondary Outcome: Percentage of Participants With Anti-Meningococcal Serogroup C (Anti-MCC) Antibody (Ab) Titre ≥1:8(1/Dil) and Titre ≥1:28 (1/Dil) One Month After Anti-Haemophilus Influenzae Type B (Anti-Hib) Vaccination (Part 2)
Description: The percentage of participants with anti-Hib Ab titres ≥1:8 (1/dil) and ≥1:28 (1/dil) were determined prior to, and 1 month after, administration of the single HiB-MCC vaccine at 12 months of age. Serum Ab levels were assayed using the Meningo C rabbit complement serum bactericidal Ab (rSBA) assay.
Time Frame: Month 12 and Month 13 (Prior to anti-Hib MCC and 1 month after anti-HiB MCC)
Population: All randomized and treated participants with data available, who had no protocol violations that could interfere with results, and received all Part 1 vaccinations are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 111 | 111
Percentage of Participants
  Pre-Hib anti-MCC: % with titre ≥1:8 (1/dil): number analyzed (Participants) | 89 | 94
  Pre-Hib anti-MCC: % with titre ≥1:8 (1/dil) | 83.1 [73.7 to 90.2] | 40.4 [30.4 to 51.0]
  Pre-Hib anti-MCC: % with titre ≥1:28 (1/dil): number analyzed (Participants) | 89 | 94
  Pre-Hib anti-MCC: % with titre ≥1:28 (1/dil) | 40.4 [30.2 to 51.4] | 16.0 [9.2 to 25.0]
  Post-Hib anti-MCC: % with titre ≥1:8 (1/dil) | 100.0 [96.7 to 100.0] | 97.3 [92.2 to 99.4]
  Post-Hib anti-MCC: % with titre ≥1:28 (1/dil) | 99.1 [95.0 to 100.0] | 95.5 [89.7 to 98.5]

16. Secondary Outcome: Antibody (Ab) Geometric Mean Titres (GMTs) for Meningococcal Serogroup C (MCC) One Month After Anti-Haemophilus Influenzae Type B (Anti-Hib) Meningococcal Serogroup C (MCC) Vaccination (Part 2)
Description: Antibody GMTs were were determined prior to, and 1 month after, administration of the single HiB-MCC vaccine at 12 months of age. Serum Ab levels were assayed using the Meningo C rabbit complement serum bactericidal Ab (rSBA) assay.
Time Frame: Month 12 and Month 13 (Prior to anti-Hib MCC and 1 month after anti-HiB MCC)
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: tire (1/dil)
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 111 | 111
tire (1/dil)
  Pre-Hib anti-MCC GMT: number analyzed (Participants) | 89 | 94
  Pre-Hib anti-MCC GMT | 50.3 [34.4 to 73.4] | 8.7 [5.9 to 12.9]
  Post-Hib anti-MCC GMT | 3257.9 [2597.4 to 4086.3] | 580.8 [432.7 to 779.5]

17. Secondary Outcome: Percentage of Participants With Anti-Polyribosylribitol Phosphate (PRP) Antibody (Ab) Titres ≥0.15 µg/mL and ≥1.0 µg/mL One Month After Anti-Haemophilus Influenzae Type B MCC Vaccination (Part 2)
Description: The percentage of participants with anti-PRP Ab titres ≥0.15 µg/mL and ≥1.0 µg/mL was determined prior to, and 1 month after, administration of the anti-Hib vaccination at Month 12. Anti-PRP Ab titres were measured with radioimmunoassay (RIA).
Time Frame: Month 4 and Month 5 (1 month after MCC-TT/MCC-CRM Doses 1 and 2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 111 | 111
Percentage of Participants
  Pre-Hib-MCC anti-PRP ≥0.15 µg/mL: number analyzed (Participants) | 82 | 87
  Pre-Hib-MCC anti-PRP ≥0.15 µg/mL | 93.9 [86.3 to 98.0] | 95.4 [88.6 to 98.7]
  Pre-Hib-MCC anti-PRP ≥1.0 µg/mL: number analyzed (Participants) | 82 | 87
  Pre-Hib-MCC anti-PRP ≥1.0 µg/mL | 54.9 [43.5 to 65.9] | 56.3 [45.3 to 66.9]
  Post-Hib-MCC anti-PRP ≥0.15 µg/mL | 100.0 [96.7 to 100.0] | 100.0 [96.6 to 100.0]
  Post-Hib-MCC anti-PRP ≥1.0 µg/mL | 99.1 [95.0 to 100.0] | 100.0 [96.6 to 100.0]

18. Secondary Outcome: Geometric Mean Titres (GMTs) for Anti-Polyribosylribitol Phosphate (PRP) Antibody (Ab) One Month After Anti-Haemophilus Influenzae Type B (HiB) MCC Vaccination (Part 2)
Description: Anti-PRP Ab GMTs were determined prior to, and 1 month after, administration of the anti-Hib vaccination at Month 12. Anti-PRP Ab titres were measured with radioimmunoassay (RIA) and are expressed as µg/mL..
Time Frame: Month 4 and Month 5 (1 month after MCC-TT/MCC-CRM Doses 1 and 2)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 111 | 111
µg/mL
  Pre-Hib-MCC anti-PRP ≥0.15 µg/mL: number analyzed (Participants) | 82 | 87
  Pre-Hib-MCC anti-PRP ≥0.15 µg/mL | 1.09 [0.81 to 1.45] | 1.18 [0.90 to 1.55]
  Pre-Hib-MCC anti-PRP ≥1.0 µg/mL: number analyzed (Participants) | 110 | 106
  Pre-Hib-MCC anti-PRP ≥1.0 µg/mL | 100.19 [81.05 to 123.86] | 121.00 [101.11 to 144.80]

19. Secondary Outcome: Percentage of Participants Experiencing an Adverse Event (AE) [Part 1]
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the investigational product, whether or not considered related to the use of the product.
Time Frame: Up to 4.5 months (up to 15 days after the final Part 1 vaccination)
Population: All randomized participants who received ≥1 dose of study medication in Part 1 are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 142 | 142
Percentage of Participants | 98.6 [95.0 to 99.8] | 97.2 [92.9 to 99.2]

20. Secondary Outcome: Percentage of Participants Experiencing an Injection Site (Vaccine-Related) Systemic Adverse Event (AE) [Part 1]
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the investigational product, whether or not considered related to the use of the product. As per protocol, all injection site AEs were considered vaccine-related.
Time Frame: Up to 4.5 months (up to 15 days after the final Part 1 vaccination)
Population: All randomized participants who received ≥1 dose of study medication in Part 1 are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 142 | 142
Percentage of Participants | 98.6 [95.0 to 99.8] | 96.5 [92.0 to 98.8]

21. Secondary Outcome: Percentage of Participants Experiencing a Solicited Injection Site Reaction (ISR) at the V419 Injection Site (Part 1)
Description: The percentage of participants with solicited ISRs was determined for each arm. Solicited ISRs consisted of injection site pain, erythema, and swelling.
Time Frame: Up to 4.5 months (up to 15 days after the final Part 1 vaccination)
Population: All randomized participants who received ≥1 dose of study medication in Part 1 are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 142 | 142
Percentage of Participants
  Erythema | 71.1 [62.9 to 78.4] | 64.8 [56.3 to 72.6]
  Pain | 63.4 [54.9 to 71.3] | 66.2 [57.8 to 73.9]
  Swelling | 51.4 [42.9 to 59.9] | 47.2 [38.8 to 55.7]

22. Secondary Outcome: Percentage of Participants Experiencing an Unsolicited Injection Site Reaction (ISR) at the V419 Injection Site (Part 1)
Description: The percentage of participants with unsolicited ISRs was determined for each arm. Unsolicited ISRs were any injection-site ISRs not considered solicited.
Time Frame: Up to 4.5 months (up to 15 days after the final Part 1 vaccination)
Population: All randomized participants who received ≥1 dose of study medication in Part 1 are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 142 | 142
Percentage of Participants | 6.3 [2.9 to 11.7] | 11.3 [6.6 to 17.7]

23. Secondary Outcome: Percentage of Participants Experiencing a Solicited Injection Site Reaction (ISR) at the MCC-TT or MCC-CRM Injection Site (Part 1)
Description: as for outcome 21
Time Frame: Up to 4.5 months (up to 15 days after the final Part 1 vaccination)
Population: All randomized participants who received ≥1 dose of study medication in Part 1 are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 142 | 142
Percentage of Participants
  Erythema | 56.3 [47.8 to 64.6] | 45.8 [37.4 to 54.3]
  Pain | 41.5 [33.3 to 50.1] | 45.8 [37.4 to 54.3]
  Swelling | 35.9 [28.0 to 44.4] | 28.2 [20.9 to 36.3]

24. Secondary Outcome: Percentage of Participants Experiencing an Unsolicited Injection Site Reaction (ISR) at the MCC-TT or MCC-CRM Injection Site (Part 1)
Description: The percentage of participants with unsolicited ISRs was determined for each arm. Unsolicited ISRs consisted of bruising, dermatitis, erythema, induration, mass, pain, rash, and warmth.
Time Frame: Up to 4.5 months (up to 15 days after the final Part 1 vaccination)
Population: All randomized participants who received ≥1 dose of study medication in Part 1 are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 142 | 142
Percentage of Participants
  Bruising | 1.4 | 4.2
  Dermatitis | 0 | 0.7
  Erythema | 0 | 0.7
  Induration | 1.4 | 0.7
  Mass | 3.5 | 2.1
  Pain | 0 | 0.7
  Rash | 1.4 | 0.7
  Warmth | 0 | 2.1

25. Secondary Outcome: Percentage of Participants Experiencing a Solicited Systemic Adverse Event (AE) [Part 1]
Description: The percentage of participants with solicited systemic AEs was determined for each arm. Solicited systemic AEs consisted of crying, decreased appetite, irritability, pyrexia, somnolence, and vomiting.
Time Frame: Up to 4.5 months (up to 15 days after the final Part 1 vaccination)
Population: All randomized participants who received ≥1 dose of study medication in Part 1 are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 142 | 142
Percentage of Participants
  Crying | 85.9 | 81.0
  Decreased appetite | 63.4 | 64.8
  Irritability | 88.0 | 81.0
  Pyrexia | 11.3 | 10.6
  Somnolence | 81.7 | 78.9
  Vomiting | 40.1 | 49.3

26. Secondary Outcome: Percentage of Participants Experiencing Increased Temperature [Part 1]
Description: The percentage of participants experiencing temperatures ≥38.0° Celsius (C), >38.5° C, and >39.5° C following any Part 1 vaccination was determined.
Time Frame: Up to 4.5 months (up to 15 days after the final Part 1 vaccination)
Population: All randomized participants who received ≥1 dose of study medication in Part 1 are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 142 | 142
Percentage of Participants
  % ≥38.0° C | 11.3 | 10.6
  % >38.5° C | 1.4 | 2.1
  % >39.5° C | 0.0 | 0.0

27. Secondary Outcome: Percentage of Participants Experiencing a Serious Adverse Event (SAE) [Part 1]
Description: An SAE is an event that results in death; is life-threatening; results in or prolongs hospitalization; is a congenital anomaly/birth defect; is a cancer; is an overdose; or is another important medical event that may jeopardize the participant.
Time Frame: Up to 4.5 months (up to 15 days after the final Part 1 vaccination)
Population: All randomized participants who received ≥1 dose of study medication in Part 1 are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
Number analyzed (Participants) | 142 | 142
Percentage of Participants | 4.2 [1.6 to 9.0] | 2.8 [0.8 to 7.1]

ADVERSE EVENTS:
Time Frame: Up to 12.5 months (up to 14 days after the final dose of study medication)
Description: All participants who received ≥1 dose of study medication are included.
Arm/Group | V419 and MCC-TT | V419 and MCC-CRM
All-Cause Mortality (participants affected / at risk) | 0/142 | 0/142
Serious Adverse Events (participants affected / at risk) | 6/142 | 4/142
Other Adverse Events (participants affected / at risk) | 140/142 | 137/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V419 and MCC-TT (N=142) | V419 and MCC-CRM (N=142)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crying (General disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis neonatal (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Weight gain poor (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V419 and MCC-TT (N=142) | V419 and MCC-CRM (N=142)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (5)
Diarrhoea (Gastrointestinal disorders) | 11 (15) | 8 (11)
Teething (Gastrointestinal disorders) | 7 (8) | 1 (1)
Vomiting (Gastrointestinal disorders) | 57 (93) | 71 (112)
Crying (General disorders) | 122 (273) | 115 (262)
Injection site bruising (General disorders) | 4 (4) | 7 (12)
Injection site erythema (General disorders) | 104 (342) | 96 (305)
Injection site mass (General disorders) | 5 (5) | 3 (4)
Injection site pain (General disorders) | 93 (258) | 100 (267)
Injection site swelling (General disorders) | 78 (211) | 70 (177)
Injection site warmth (General disorders) | 0 (0) | 3 (4)
Irritability (General disorders) | 125 (301) | 115 (286)
Pyrexia (General disorders) | 19 (22) | 18 (23)
Nasopharyngitis (Infections and infestations) | 11 (12) | 12 (14)
Rhinitis (Infections and infestations) | 8 (8) | 6 (7)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 91 (164) | 92 (167)
Somnolence (Nervous system disorders) | 116 (227) | 112 (231)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 6 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No